CLINICAL TRIAL: NCT02874222
Title: E1Z11 A Cohort Study to Evaluate Genetic Predictors of Aromatase Inhibitor, AIMSS
Brief Title: A Cohort Study to Evaluate Genetic Predictors of Aromatase Inhibitor Musculoskeletal Symptoms
Acronym: AIMSS
Status: Completed | Type: Observational
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: Alliance for Clinical Trials in Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: NMCSD.2014.0053
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
Keywords: aromatase inhibitors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Caucasian: surveys completed by subject n=600, nationally
  Interventions: Other: surveys completed by subject
- African-American: surveys completed by subject n=200, nationally
  Interventions: Other: surveys completed by subject
- Asian: surveys completed by subject n=200, nationally
  Interventions: Other: surveys completed by subject

INTERVENTIONS:
Other: surveys completed by subject — Cohort study designed to validate previously identified associations between 10 specific SNPs and discontinuation of treatment with AIs due to the development of MSS among women with breast cancer.

SUMMARY:
Breast cancer is one of the most prevalent cancers with 207,090 new cases of breast cancer and 39,840 deaths in women predicted for 2010 in the United States. Aromatase inhibitors (AIs) are used as first-line adjuvant therapy for postmenopausal women with early stage breast cancer. The effectiveness of current therapy is widely recognized to be compromised by poor compliance because of aromatase inhibitor-associated musculoskeletal symptoms (AIMSS), a syndrome that affects up to 40-50% of women who take these medications. The syndrome that was not recognized during the registration trials for this class of drugs, it can lead to discontinuation in up to 24% of women over 2 years. Knowledge that can be used to prevent discontinuation of these important agents because of severe AIMSS is urgently needed.

DETAILED DESCRIPTION:
The NCI Division of Cancer Prevention has recognized AIMSS as a priority area for future study. The symptoms are associated with a high rate of AI discontinuation and therefore compromise survival outcomes at great cost to both patients and society. Very little is known about AIMSS, or how to predict who is at risk for the condition, or for discontinuing therapy because of the symptoms. This study will provide a basis for comprehensive assessment of risk factors at the patient-reported outcomes, phenotypic, and laboratory levels. We will explore the natural history of AIMSS in different ethnic populations, and will validate previously reported genetic determinants of the development of AIMSS. A common problem with multicenter GWAS studies of very large sample size, especially in the absence of measurable diagnostic parameters, is inclusion of heterogeneous groups of patients. In addition to assessing pharmacogenomic predictors, this study involves specification of a pre-defined AIMSS phenotype and collection of patient-reported outcomes (PROs). As such, these data will have clinical utility by clarifying the factors associated with aromatase inhibitor discontinuation and thus guiding clinicians towards interventions to improve adherence. Coupled with other studies, the long-term goals are to develop a gene signature that will be used to better guide the selection of endocrine interventions for patients with breast cancer. The underlying physiology of AIMSS remains obscure. A small exploratory case control study did not find a role for commonly encountered cytokines in AIMSS. The role of estrogen and estrogen metabolites remains a possible explanatory variable, as well as new cytokines such as IL-17. This newly described cytokine has been implicated in disorders such as rheumatoid arthritis and other autoimmune diseases, and has been specifically linked to articular nociception in animal models of arthritis. AIMSS Phenotype: The large studies to date of AIs (ATAC, BIG I-98, E1Z03) have been limited by the absence of a clearly defined phenotype for AIMSS. Retrospective analyses have provided some information that clearly cannot replace (PROs). The lack of good prospective PROs represents a major gap as a well-defined phenotype is necessary in order to identify useful genomic associations. Methods evaluating possible predictors such as the use of MRI of the wrists for tenosynovitis are expensive and have not been definitive, and patient-reported symptoms are used and may represent the most useful clinical phenotype.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 60 years of age; or
* < 60 years of age and amenorrheic for ≥ 12 months prior to day 1 if uterus/ovaries are intact; or
* < 60 years of age, and the last menstrual period 6-12 months prior to day 1, if intact uterus/ovaries and meets biochemical criteria for menopause (FSH and estradiol within institutional standard for postmenopausal status); or
* < 60 years of age, without a uterus, and meets biochemical criteria for menopause (FSH and estradiol within institutional standards for postmenopausal status); or
* < 60 years of age and history of bilateral oophorectomy. Surgery must have been completed at least 4 weeks prior to day 1; or
* Prior radiation castration with amenorrhea for at least 6 months.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: breast cancer patients
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2023-07 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
development of arthritic symptoms | 12 months
  patients surveyed and given physical exams

CONTACTS AND LOCATIONS:
Overall Officials: Preston Gable, MD, Principal Investigator — Site PI
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes